CLINICAL TRIAL: NCT06640036
Title: FILIP: Fat Intake, Inflammation and LIPids
Acronym: FILIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Chalmers University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-03117-01
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-04

CONDITIONS: Cardiometabolic Risk Factors; Inflammation; Microbiota
Keywords: Blood lipid profile; Low grade inflammation
MeSH Terms: conditions — Inflammation | interventions — Rapeseed Oil; Butter; Coconut Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Meals identical in apperance and taste will be prepared, and blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1: Rapeseed oil, butter, coconut oil (Experimental): Diets rich in rapeseed oil, butter or coconut oil given in blinded, preprepared meals
  Interventions: Other: Rapeseed oil; Other: Butter; Other: Coconut oil
- Sequence 2: Rapeseed oil, coconut oil, butter (Experimental): Diets rich in rapeseed oil, butter or coconut oil given in blinded, preprepared meals
  Interventions: Other: Rapeseed oil; Other: Butter; Other: Coconut oil
- Sequence 3: Butter, coconut oil , rapeseed oil (Experimental): Diets rich in rapeseed oil, butter or coconut oil given in blinded, preprepared meals
  Interventions: Other: Rapeseed oil; Other: Butter; Other: Coconut oil
- Sequence 4: Butter, rapeseed oil, coconut oil (Experimental): Diets rich in rapeseed oil, butter or coconut oil given in blinded, preprepared meals
  Interventions: Other: Rapeseed oil; Other: Butter; Other: Coconut oil
- Sequence 5: Coconut oil, rapeseed oil, butter (Experimental): Diets rich in rapeseed oil, butter or coconut oil given in blinded, preprepared meals
  Interventions: Other: Rapeseed oil; Other: Butter; Other: Coconut oil
- Sequence 6: Coconut oil, butter, rapeseed oil (Experimental): Diets rich in rapeseed oil, butter or coconut oil given in blinded, preprepared meals
  Interventions: Other: Rapeseed oil; Other: Butter; Other: Coconut oil

INTERVENTIONS:
Other: Rapeseed oil — During 1 week, 46 % of total energy intake will come from rapeseed oil, using pre-prepared and blinded meals.
Other: Butter — During 1 week, 46 % of total energy intake will come from butter, using pre-prepared and blinded meals.
Other: Coconut oil — During 1 week, 46 % of total energy intake will come from coconut oil, using pre-prepared and blinded meals.

SUMMARY:
Low-grade inflammation is involved in the pathogenesis of type 2 diabetes and cardiovascular disease. Increasing evidence suggests that dietary intake may be involved in the inflammatory process. How nutritional composition of the diet affects the inflammatory response is however not well understood.

The aim of this project is to study if intake of three different fat sources induce different effects on inflammation markers, blood lipids, blood glucose and the microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Willing to eat the study diet

Exclusion Criteria:

* malabsorption-related condition
* contraindications to consume a high fat diet
* intolerance to any foods used in the study (e.g. cow's milk, egg, gluten)
* established cardiovascular disease, diabetes or cancer
* current use of medication known to affect lipid metabolism (e.g. statins) or inflammation (e.g. NSAID, glucocorticoids).
* hemoglobin <100 g/L
* ongoing pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Total cholesterol | Baseline and 1 week
hs-CRP | Baseline and 1 week
  High sensitivity C-reactive Protein

SECONDARY OUTCOMES:
Inflammation markers | Baseline and 1 week
  Eg. GlycA, IL6, TNF-a
Blood lipid propfile | Baseline and 1 week
  Blood lipids and their subfractions, lipoproteins, apolipoproteins
Glucose | Continuous during 1 week
  Glucose, measured by continuous blood glucose monitoring
Microbiota | Baseline and 1 week
  Change in gut microbial composition and diversity (alpha- and beta).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
It would depend on ethical permission to share the IPD.